CLINICAL TRIAL: NCT03875027
Title: Outcome of Proximal Femur Replacement at a Tertiary Care Hospital
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, shah fahad, RESIDENT, Aga Khan University
Other Study IDs: akupd
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Outcome, Fatal
Keywords: proximal femur; functional outcome; fracture; failed hip surgery
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: proximal femur replacement — patient with proximal femur fracture or those in whom previous surgery on hip is failed and treated with replacement of proximal femur implant

SUMMARY:
This is a retrospective review of all patients who underwent PFR for either bipolar hemiarthroplasty or total hip replacement

DETAILED DESCRIPTION:
retrospective review of all patients who underwent PFR for either bipolar hemiarthroplasty or total hip replacement will be conducted All patients that fall in the selection criteria from 2009 to 2018 will be included as part of this study will be selected Patients are identified using medical record numbers. A questionnaire containing questions on demographics of the patients which includes their age, sex and co morbids. Furthermore, the cause of fracture, time from the fracture to presentation in the emergency room, time from the presentation to ER to the time patient was in the operating room would be noted. Duration of the surgery.

The weight bearing status in the ward and follow-up would be noted. Functionality of the patient; which is that how much patients are able to carry their normal daily routine work would also be noted from the medical records.

Collected data will be analysed using Statistical Package for Social Sciences (SPSS, Inc, Chicago, IL, USA). Results will be recorded as frequencies, means, Standard Deviation (SD) and p-values while statistical tests will be applied for comparative reasons. For all purposes a p-value of 0.05 will be considered as the level of significance.

ELIGIBILITY:
Inclusion Criteria:

* All patients, regardless of race, gender, age and co-morbids, who were treated with proximal femur fracture with any of the following variables:

Poor bone quality Bone loss Severe communition Multiple comorbids Failed hip surgery Pathological fractures

Exclusion Criteria:

* The patient who weren't treated with proximal femoral replacemnt, those lost to follow up, those with missing record.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient underwent proximal femur replacement
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
functional outcome | 2009 till 2018
  improvement in functional claculated via harris hip score

SECONDARY OUTCOMES:
mortality | one year
  death within one of year of surgery

IPD SHARING:
Plan to Share IPD: Undecided